CLINICAL TRIAL: NCT00383916
Title: An Open-Label, Single-Dose, Randomized, 2-Period, Crossover, Bioequivalence Study Between the Altana Formulation of Pantoprazole Delayed-Release Granules and the Wyeth Formulation of Pantoprazole Delayed-Release Granules in Healthy Subjects.
Brief Title: Study Comparing 2 Different Formulations of Pantoprazole in Healthy Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3001B1-119
Record Dates: First submitted 2006-10-02; First posted 2006-10-04 (Estimated); Last update posted 2007-03-08 (Estimated); Status verified 2007-03

CONDITIONS: Healthy Subjects
Keywords: healthy
MeSH Terms: interventions — Pantoprazole

INTERVENTIONS:
Drug: pantoprazole

SUMMARY:
A study comparing 2 different investigational formulations of pantoprazole in healthy adults.

DETAILED DESCRIPTION:
open-label, single-dose, randomized, 2-period, 2-sequence, crossover, inpatient bioequivalence study

ELIGIBILITY:
Inclusion Criteria

* Men or women aged 18 to 50 years.
* Healthy as determined by the investigator.

Exclusion Criteria

* History or active presence of clinically important medical disease.
* History of drug or alcohol abuse.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2006-10; Study Completion 2006-10

PRIMARY OUTCOMES:
To determine the bioequivalence of the Altana formulation of pantoprazole to the Wyeth formulation of pantoprazole delayed-release granules.

SECONDARY OUTCOMES:
To obtain additional safety and tolerability data concerning pantoprazole in healthy subjects and to assess the pharmacokinetics of the Altana formulation.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer